CLINICAL TRIAL: NCT05980780
Title: Video Developed for Children With Familial Mediterranean Fever The Effect of Game on Disease Management and Quality of Life
Brief Title: The Effect of Video Game on Children With Familial Mediterranean Fever
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gamze Kas Alay, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-KAEK-7
Record Dates: First submitted 2023-07-21; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: FMF
Keywords: child; mobile game; disease management; quality of life; disease education

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Masking will be used when making the statistical evaluation of the results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The control group (No Intervention): no intervention
- video game group (Experimental): Children in this group will play a video game for disease management
  Interventions: Behavioral: video game group
- Education booklet group (Experimental): Children in this group will read an educational booklet for disease management.
  Interventions: Behavioral: Education booklet group

INTERVENTIONS:
Behavioral: video game group — Pretest: Participants will be informed about FMF, treatment of FMF, side effects of treatment, factors that trigger attacks, symptoms that occur during the attack, symptom management/disease self-management, and coping with stress through a video game. At the beginning of the application, questions for the collection of demographic data and scales applied to the control group will be applied. The game will be played at home once a week for 1 month. For this, reminder messages will be sent once a week by obtaining the contact information of the mothers.
  Post-test 1: The scales will be re-administered 1 month after the pre-test. Post-test 2: The scales will be administered again 3 months after the pre-test.
  Arms: video game group
Behavioral: Education booklet group — Pretest: Participants will be informed about FMF, treatment of FMF, side effects of treatment, factors that trigger attacks, symptoms that occur during the attack, symptom management/disease self-management, and coping with stress through a training booklet. At the beginning of the application, questions for the collection of demographic data and scales applied to the control group will be applied. The booklet will be read at home once a week for 1 month. For this, reminder messages will be sent once a week by obtaining the contact information of the mothers.
  Post-test 1: The scales will be re-administered 1 month after the pre-test. Post-test 2: The scales will be administered again 3 months after the pre-test.
  Arms: Education booklet group

SUMMARY:
This study was planned to be carried out as a pretest-posttest control group design in experimental type and randomized groups in order to determine the effect of educating children aged 8-14 with a diagnosis of Familial Mediterranean Fever through a mobile game application and training booklet on their disease knowledge, disease self-efficacy, symptom management and quality of life.

H0: Informing children with Familial Mediterranean Fever through mobile games and educational booklets has no effect on the child's knowledge of the disease, disease self-efficacy, symptom management and quality of life.

Compared to children with Familial Mediterranean Fever who were informed by mobile games, and children with Familial Mediterranean Fever who were informed through the education booklet and were not informed at all; H1: Disease knowledge increases. H2: Disease self-efficacy increases. H3: The number of attacks, activity intolerance, number of symptoms and severity of pain decrease.

H4: Quality of life increases.

DETAILED DESCRIPTION:
Today, with the ease of access to technological tools, the use of mobile technologies by children, adolescents and health professionals is becoming increasingly common. These technologies have begun to change the way healthcare professionals provide healthcare services, and support children's participation in their own care by providing easy-to-use digital services. It is emphasized that these technologies, which are accepted with interest by children and young people, are important new tools in providing health-related behavior change in children. One of these channels is video games developed for health. The use of video games in education as a method of children's choice is an important channel that will enable them to feel that they are in control of their own lives at an earlier age. Thus, these alternative education methods for children and adolescents can make a difference in patient education and management of chronic diseases. In the literature, it has been shown that video games are used and effective in psychotherapy practices and oral and dental health education, especially in the management of chronic diseases such as diabetes, cancer and asthma. However, no study has been found on disease self-management and education in children for Familial Mediterranean Fever, which is very common in our country and continues throughout life. We think that under the control of Familial Mediterranean Fever, which is a chronic disease, the child's self-management will manage the disease better, the frequency of attacks and hospital admissions will decrease, and future complications can be prevented.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with FMF (early 1 month)
* Taking colchicine medication
* Having an attack at least once a year
* Willingness to participate in the research
* His family's consent to participate in the research
* Being literate

Exclusion Criteria:

* Any identified mental disability
* Speech and communication difficulties

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Disease self-efficacy Self-Efficacy Scale for Pediatric Chronic Disease | before the intervention, immediately after the intervention, 2 months after the intervention
  The Pediatric Self-Efficacy Scale for Chronic Disease (PRCISE) is an 11-point Likert-type scale consisting of 15 all positive items. The score of each item in the scale ranges from 0 to 10 and consists of statements such as "not sure at all" for 0 and "very sure" for 10. The scale, in which the level of self-efficacy increases as the score increases, is evaluated over 150 points.
Life quality | before the intervention, immediately after the intervention, 2 months after the intervention
  A Multi-Dimensional Assessment Scale for Children with Autoinflammatory Disease (JAIMAR) consists of 16 items in total, including assessment of functional skills, pain, compliance with drug use, and quality of life. The measure of quality of life; physical status, social status, school status and emotional status sub-dimensions are available. In addition, the form includes descriptive questions to be used in patient follow-up. In the scale scoring, 5-point Likert-type rating (Never=1, Rarely=2, Sometimes=3, Frequently=4, Always=5) is used in the sub-dimensions of quality of life (physical, social, school and emotional state), and the scoring is 1 It is done from th to 5th. After the average of the answers given to the questions in the criterion is taken, it is rescaled so that the highest score is 10. The quality of life criterion is calculated in the same way by using the average of the questions in all sub-criteria.
Disease information | before the intervention, immediately after the intervention, 2 months after the intervention
  It is a short knowledge test of 11 questions, which was created by researchers and aims to measure disease knowledge. The questions in the test are closed-ended as yes/no, and the child who ticks yes is asked to write an explanation in the adjacent box.

CONTACTS AND LOCATIONS:
Overall Officials: Birsen MUTLU, Phd, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sparapani VC, Fels S, Kamal N, Ortiz La Banca R, Nascimento LC. A Video Game for Brazilian T1D Children about Knowledge of Disease and Self-care: A Methodological Study. J Diabetes Sci Technol. 2022 Nov;16(6):1444-1450. doi: 10.1177/19322968211017555. Epub 2021 May 28. PMID 34044626
- [Background] Rafeezadeh, E., Ghaemi, N., Miri, H.H., Rezaeian, A., (2019). Effect of an Educational Video Game for Diabetes Self-management on Adherence to a Self-care Regimen in Children with Type 1 Diabetes. Evidence Based Care Journal, 9 (1), 74-83.
- [Background] Nascimento Lda S, de Gutierrez MG, De Domenico EB. [Educative programs based on self-management: an integrative review]. Rev Gaucha Enferm. 2010 Jun;31(2):375-82. doi: 10.1590/s1983-14472010000200024. Portuguese. PMID 21500520
- [Background] Migita K, Asano T, Sato S, Koga T, Fujita Y, Kawakami A. Familial Mediterranean fever: overview of pathogenesis, clinical features and management. Immunol Med. 2018 Jun;41(2):55-61. doi: 10.1080/13497413.2018.1481579. Epub 2018 Sep 7. PMID 30938266
- [Background] Hentgen V, Grateau G, Kone-Paut I, Livneh A, Padeh S, Rozenbaum M, Amselem S, Gershoni-Baruch R, Touitou I, Ben-Chetrit E. Evidence-based recommendations for the practical management of Familial Mediterranean Fever. Semin Arthritis Rheum. 2013 Dec;43(3):387-91. doi: 10.1016/j.semarthrit.2013.04.011. Epub 2013 Jun 3. PMID 23742958
- [Background] Yildirim DG, Bakkaloglu SA, Acar ASS, Celik B, Buyan N. Evaluation of quality of life and its associations with clinical parameters in pediatric patients with familial Mediterranean fever. North Clin Istanb. 2021 Apr 26;8(3):255-260. doi: 10.14744/nci.2020.90093. eCollection 2021. PMID 34222806
- [Background] Gezgin Yildirim D, Gonen S, Fidan K, Soylemezoglu O. Does Age at Onset Affect the Clinical Presentation of Familial Mediterranean Fever in Children? J Clin Rheumatol. 2022 Jan 1;28(1):e125-e128. doi: 10.1097/RHU.0000000000001637. PMID 33252389
- [Background] Yildirim DG, Bakkaloglu SA, Soysal-Acar AS, Buyan N. Parental knowledge about familial Mediterranean fever: a cross-sectional study. Turk J Pediatr. 2021;63(6):1048-1055. doi: 10.24953/turkjped.2021.06.013. PMID 35023655
- [Background] Durmuş, S.Y., Ozlu, S.G., Cop, E., Bulbul, M. (2022). Health Related Quality of Life of Children Aged 2-18 Years with Familial Mediterranean Fever. Turkish Journal of Pediatric Disease, Elektronik yayın tarihi 24.02.2022 DOI: 10.12956/tchd.1013742
- [Background] Charlier N, Zupancic N, Fieuws S, Denhaerynck K, Zaman B, Moons P. Serious games for improving knowledge and self-management in young people with chronic conditions: a systematic review and meta-analysis. J Am Med Inform Assoc. 2016 Jan;23(1):230-9. doi: 10.1093/jamia/ocv100. Epub 2015 Jul 17. PMID 26186934
- [Background] Calle-Bustos AM, Juan MC, Garcia-Garcia I, Abad F. An augmented reality game to support therapeutic education for children with diabetes. PLoS One. 2017 Sep 28;12(9):e0184645. doi: 10.1371/journal.pone.0184645. eCollection 2017. PMID 28957355
- [Background] Bravo L, Killela MK, Reyes BL, Santos KMB, Torres V, Huang CC, Jacob E. Self-Management, Self-Efficacy, and Health-Related Quality of Life in Children With Chronic Illness and Medical Complexity. J Pediatr Health Care. 2020 Jul-Aug;34(4):304-314. doi: 10.1016/j.pedhc.2019.11.009. Epub 2020 Feb 25. PMID 32107073
- [Background] Baranowski T, Buday R, Thompson DI, Baranowski J. Playing for real: video games and stories for health-related behavior change. Am J Prev Med. 2008 Jan;34(1):74-82. doi: 10.1016/j.amepre.2007.09.027. PMID 18083454